CLINICAL TRIAL: NCT02700165
Title: Non-Invasive Fat Reduction in the Chin Using Cryolipolysis
Brief Title: Fat Reduction in the Submandibular/Submental Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA15-006
Record Dates: First submitted 2016-01-28; First posted 2016-03-07 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-05

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- CoolSculpting with CoolMini (Experimental): The treatments are designed to see if fat in the submandibular/submental area (chin), can be reduced using cryolipolysis.
  Interventions: Device: The ZELTIQ CoolSculpting System

INTERVENTIONS:
Device: The ZELTIQ CoolSculpting System — The CoolSculpting device will be used to perform the treatments.

SUMMARY:
The purpose of this study is to further evaluate the safety and efficacy of non-invasive reduction of subcutaneous fat in the submental and submandibular area using Cryolipolysis.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 22 years of age and < 65 years of age.
* Submental and submandibular skin fold thickness > 1cm (measured by caliper).
* No weight change exceeding 5% of body weight in the preceding month.
* Agreement to maintain his/her weight (i.e., within 5%) by not making any major changes in diet or exercise routine during the course of the study.
* Subject has signed a written informed consent form.

Exclusion Criteria

* Skin laxity in the neck or chin area for which reduction in submental and submandibular fat may, in the opinion of the investigator, result in an unacceptable aesthetic result.
* Prominent platysmal bands at rest which may interfere with assessment of submental fat
* Evidence of any cause of enlargement in the submental area other than localized subcutaneous fat, such as swollen lymph nodes or ptotic submandibular glands.
* Significant enlargement on the anterior neck that may prevent the proper placement of the applicator e.g. enlarged thyroid glands.
* Treatment with dermal fillers, radiofrequency or laser procedures, or chemical peels in the neck or chin area (below the mandible) within the past 6 months.
* Botulinum toxin or other aesthetic drug injections within the neck or chin area (below the mandible) within the past 6 months.
* History of facial nerve paresis or paralysis (such as Bell's palsy).
* History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.) or implant in or adjacent to the area of intended treatment.
* History of prior neck surgery, or prior surgery in the area of intended treatment.
* Current dental infection.
* Known history of cryoglobulinemia, cold urticaria, cold agglutinin disease or paroxysmal cold hemoglobinuria.
* Known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Currently taking or has taken diet pills or weight control supplements within the past month.
* Any dermatological conditions, such as scars in the location of the treatment area that may interfere with the treatment or evaluation.
* Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Pregnant or intending to become pregnant in the next 6 months.
* Lactating or has been lactating in the past 6 months.
* Unable or unwilling to comply with the study requirements.
* Currently enrolled in a clinical study of an unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bernstein, MD, Principal Investigator — Main Line Center for Laser Surgery
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernstein EF, Bloom JD. Safety and Efficacy of Bilateral Submental Cryolipolysis With Quantified 3-Dimensional Imaging of Fat Reduction and Skin Tightening. JAMA Facial Plast Surg. 2017 Sep 1;19(5):350-357. doi: 10.1001/jamafacial.2017.0102. PMID 28426847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects seeking reduction of fat in the submental and submandibular area were recruited from the general population.
Groups:
- CoolSculpting With CoolMini Applicator for Fat Reduction in the Chin: Per protocol, subjects were permitted to receive up to 3 CoolSculpting treatments on the submental and submandibular area at each of two treatment sessions spaced 6 weeks apart. At each treatment session, subjects were treated with the CoolSculpting device programmed for a specified protocol-defined time and temperature. All subjects received 2 cooling cycles at the first treatment session. At the second treatment visit, 12 subjects received 2 cooling cycles and 2 received 1 cycle.
Period: Overall Study
Arm/Group | CoolSculpting With CoolMini Applicator for Fat Reduction in the Chin
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- CoolSculpting With CoolMini Applicator: ZELTIQ CoolSculpting System Treatment Group
Arm/Group | CoolSculpting With CoolMini Applicator
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 50.5 [27 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 2
  Asian | 0
  Caucasian | 12
  Hispanic | 0
  Other | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 33.1 [21.4 to 34.3]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Accurately Identified Pre-Treatment Photos by a Panel of Blinded Independent Reviewers
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Success is defined as 70% correct identification of pre-treatment images by at least 70% correct identification of pre-treatment images by two out of three reviewers.
Time Frame: Baseline (pre-treatment) and 12 weeks post treatment
Population: All subjects were included in the analysis population.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Arm/Group | CoolSculpting With CoolMini Applicator
Number analyzed (Participants) | 14
Number analyzed (photos) | 14
photos | 11
Statistical Analysis 1: Comparison: CoolSculpting With CoolMini Applicator; Test type: Other; sucess proportion = 78.6, 95% CI 2-sided [49.2 to 95.3] — Independent physician reviewers correctly identified 13/14, 11/14 and 10/14, respectively for an overall percentage of correct identification of 34/42 or 81%. Two of three reviewers correctly identified 11/14 (78.6%) photos

2. Primary Outcome: The Number of Unanticipated Adverse Device Effects (UADE) Reported
Description: The primary safety endpoint is the count of unanticipated adverse device effects (UADEs) reported in the study period. It is expected there will be zero UADEs.
Time Frame: Enrollment through the 12 week final follow-up visit
Population: The per-protocol population of 14 subjects was analyzed.
Measure: Number; unit: UADEs
Arm/Group | CoolSculpting With CoolMini Applicator
Number analyzed (Participants) | 14
UADEs | 0

3. Secondary Outcome: Change in Fat Layer Thickness of the Submental Area as Measured by Caliper
Description: Caliper measurements will be collected prior to treatment (pre-treatment) and at the 12-week follow-up visit. The caliper measurement process involves pinching the tissue within the treatment area in order to obtain the measurement, thereby folding the tissue and doubling the fat layer thickness. Measurements were taken with subjects standing in a neutral position.
  Measured values (mm) will be halved to reflect single fat layer change and will not take into account the fold of tissue during the measurement process. The fat layer measured pre-treatment will be compared to the 12-week post-treatment measurement.
Time Frame: Baseline and 12 week post-treatment
Measure: Mean (Standard Deviation); unit: millimeters fat layer change
Groups:
- CoolSculpting With CoolMini Applicator: The ZELTIQ CoolSculpting System Treatment Group
Arm/Group | CoolSculpting With CoolMini Applicator
Number analyzed (Participants) | 14
millimeters fat layer change | -2.3 (0.8)

4. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction as assessed by questionnaires administered at 12 weeks. Subjects will be asked to determine overall satisfaction with the treatment using a 5-point scale and free-text response options on a questionnaire. The choice options will be 1 = very dissatisfied, 2- dissatisfied, 3 - not sure, 4- satisfied and 5- very satisfied. Positive responses to questionnaire statements (score 4 or 5) will be used to assess satisfaction with the CoolSculpting procedure.
Time Frame: 12 weeks post-treatment
Population: The per-protocol population of 14 subjects was included the analysis group.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting With CoolMini Applicator
Number analyzed (Participants) | 14
Participants
  Procedure comfortable/very comfortable: number analyzed (Participants) | 13
  Procedure comfortable/very comfortable | 7
  Visible fat/very visible fat reduction | 10
  Agree/strongly agree appearance more youthful: number analyzed (Participants) | 13
  Agree/strongly agree appearance more youthful | 9
  Agree/strongly agree chin looked more toned | 12
  Agree/strongly agree less self-conscious of chin | 11
  Agree/strongly agree appearance improved | 11
  Agree/strongly agree result was as expected | 11
  Satisfied/very satisfied with CoolSculpting | 13
  Would recommend procedure to a friend | 13

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment through the 12 week final follow-up visit.
Arm/Group | CoolSculpting With CoolMini Applicator
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 3/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoolSculpting With CoolMini Applicator (N=14)
Hip Replacement (Musculoskeletal and connective tissue disorders) | 1 (1) — Hip replacement performed during study period. Unrelated to study device or procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoolSculpting With CoolMini Applicator (N=14)
Rash on face and neck (Skin and subcutaneous tissue disorders) | 1 (1) — Mild rash. Not related to device or procedure.
Ear pain (Surgical and medical procedures) | 1 (1) — Mild ear pain beginning day of treatment; resolved in 5 days. Possibly related to device or procedure.
Tongue tingling (General disorders) | 1 (1) — Mild tongue tingling resolved within 7 days. Possibly related to device or procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No